CLINICAL TRIAL: NCT05927389
Title: BONeMOVE : an Adapted Physical Activity Program (APA) for Effort Rehabilitation of Children and Teenagers With Osteogenesis Imperfecta: an Interventional, Prospective, Regional, Bicentric Study.
Brief Title: Adapted Physical Activity Program (APA) for Effort Rehabilitation of Children and Teenagers With Osteogenesis Imperfecta
Acronym: BONeMOVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RC31/23/0248
Record Dates: First submitted 2023-06-13; First posted 2023-07-03 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Osteogenesis Imperfecta
Keywords: Osteogenesis Imperfecta; Children; Adolescents; Maximum oxygen consumption; Adapted physical activity; Effort rehabilitation
MeSH Terms: conditions — Osteogenesis Imperfecta

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group: 6 months APA program (Experimental): The various assessments will be carried out during 2 visits at 6 months interval as part of the usual follow-up at the "Constitutional Bone Diseases" unit at the Toulouse University Hospital.
  The APA program built from the initial assessment will be returned to the child and his family during a videoconference.
  In addition, a regular reassessment and adjustment of this program will be made every 15 days during phone calls by the APA coach.
  Interventions: Other: Adapted Physical Activity program

INTERVENTIONS:
Other: Adapted Physical Activity program — The Adaptated Physical Activity program consists of a Personalized Training Program adapted to each patient's condition and capacities

SUMMARY:
This research study aims to evaluate the effect of a 6-month adapted physical activity program (APA) on the endurance capacities (evaluated as the maximum oxygen consumption [VO2 peak]) of children and adolescents with Osteogenesis Imperfecta.

DETAILED DESCRIPTION:
Osteogenesis Imperfecta (OI) is a rare genetic disease characterised mainly by bone fragility, decreased bone mass and a susceptibility to fractures of varying severity. Different forms have been described according to the severity of the bone manifestations. Although it is a genetically heterogeneous disease, approximately 90% of OI patients have a mutation in the gene encoding gene encoding type 1 collagen, a major component of the extracellular matrix.

Chronic fatigue and decreased physical endurance are almost constant complaints of patients with OI (more than 95% according to some studies), which impacts the activities of daily living and quality of life of these patients. The causes of this decrease in endurance are multifactorial involving prolonged immobilisation secondary to fractures, chronic osteoarticular pain, but also primary muscle damage.

Mechanography studies carried out in children with OI have shown a significant deficit in muscle function in terms of both strength and power.

In healthy adults, physical inactivity is an important predictor of feeling of tired. In addition, in some chronic diseases (such as multiple sclerosis, rheumatoid arthritis or systemic lupus erythematosus), physical activity and training have been shown to be effective in improving muscle strength and functional capacity as well as fatigue and quality of life. In OI, it has been reported that physical activity improves muscle function and bone mass. Patients with OI should therefore benefit from a regular exercise programme taking into account their risk of fracture.

This study aims to evaluate the effect of a life-skills physical activity (LSPA) programme on the endurance capacities and quality of life of children and adolescents with OI.

The VO2 peak evolution will be evaluated after 6 months of program. This is a recognized parameter for the evaluation of endurance and has been validated in children. The hypothesis of this study is that the implementation of a physical activity program adapted to the daily life and interests of the child with OI will efficiently improve endurance, prevent deconditioning and promote long term benefits.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed Osteogenesis Imperfecta
* Informed and written consent signed by at least one of the two holders of parental authority
* Patient affiliated to a social security scheme or equivalent

Exclusion Criteria:

* Non-walking children (unable to perform the effort test)
* Pregnant or breastfeeding
* Participation in other interventional research

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline maximum endurance capacity at 6 months | Change from Baseline to 6 months
  Maximum oxygen consumption (VO2 peak) during an exercise test will be measured

SECONDARY OUTCOMES:
Change from baseline quality of life questionnaire score at 6 months | Change from Baseline to 6 months
  Osteogenesis Imperfecta Specific Quality of Life Questionnaire (OIQoL). Total scores are based on a 0-100 scale, where a high score represents better quality of life
Change from baseline number of steps at 6 months | Change from Baseline to 6 months
  6-minute walk test (6MWT) assessed by connected watch
Change from baseline Weight at 6 months | Change from Baseline to 6 months
  Body Mass Index

CONTACTS AND LOCATIONS:
Overall Officials: Thomas EDOUARD, MD, Principal Investigator — University Hospital, Toulouse
Locations (2):
- France (2):
  - CHU Montpellier Hôpital Arnaud de Villeneuve, Montpellier
  - CHU Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sillence DO, Senn A, Danks DM. Genetic heterogeneity in osteogenesis imperfecta. J Med Genet. 1979 Apr;16(2):101-16. doi: 10.1136/jmg.16.2.101. PMID 458828
- [Background] Rossi V, Lee B, Marom R. Osteogenesis imperfecta: advancements in genetics and treatment. Curr Opin Pediatr. 2019 Dec;31(6):708-715. doi: 10.1097/MOP.0000000000000813. PMID 31693577
- [Background] Monti E, Mottes M, Fraschini P, Brunelli P, Forlino A, Venturi G, Doro F, Perlini S, Cavarzere P, Antoniazzi F. Current and emerging treatments for the management of osteogenesis imperfecta. Ther Clin Risk Manag. 2010 Sep 7;6:367-81. doi: 10.2147/tcrm.s5932. PMID 20856683
- [Background] Arponen H, Waltimo-Siren J, Valta H, Makitie O. Fatigue and disturbances of sleep in patients with osteogenesis imperfecta - a cross-sectional questionnaire study. BMC Musculoskelet Disord. 2018 Jan 8;19(1):3. doi: 10.1186/s12891-017-1922-5. PMID 29310646
- [Background] Harsevoort AGJ, Gooijer K, van Dijk FS, van der Grijn DAFM, Franken AAM, Dommisse AMV, Janus GJM. Fatigue in adults with Osteogenesis Imperfecta. BMC Musculoskelet Disord. 2020 Jan 3;21(1):6. doi: 10.1186/s12891-019-3000-7. PMID 31900144